CLINICAL TRIAL: NCT02886312
Title: Evaluation of Oxygen Delivery Through Nasal Cannula in Volunteers
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: IRB_00083180
Record Dates: First submitted 2016-08-19; First posted 2016-09-01 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2017-12

CONDITIONS: Oxygen Delivery; Patient Monitoring; Patient Comfort

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Supplemental Oxygen Delivery System

SUMMARY:
This study will evaluate patient comfort and oxygen delivery efficiency when providing supplemental oxygen through a nasal cannula to volunteers using an instrumented oxygen delivery system. The goals of the study are to evaluate different oxygen flow rates and oxygen delivery modes. In addition, the investigators will investigate if the system can detect apnea (cessation of breathing) and removal of the nasal cannula. The investigators will also investigate how well high flow oxygen delivered only during inspiration is tolerated and how much the end-tidal oxygen increases after two minutes of high oxygen flow delivered only during the inhalation phase of the breath.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers drawn from the general public and students, staff, and faculty of the University of Utah.

Exclusion Criteria:

* Volunteers who self report respiratory diseases such as acute respiratory distress syndrome, pneumonia and lung cancer will be excluded. In addition, volunteers who self report respiratory conditions such as nasal or bronchial congestion due to a cold or allergies will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers drawn from the general public and students, staff, and faculty of the University of Utah.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
End-tidal Oxygen | Continuously throughout 30 minute volunteer study
  Did the novel system increase end-tidal oxygen?
Patient Comfort | Every 2 minutes up to 30 minutes
  Did the patients feel it was more comfortable for a given end-tidal oxygen level?
End-tidal Carbon Dioxide | Continuously throughout 30 minute volunteer study
  Was end-tidal carbon dioxide measured more accurately using the novel system?
Respiratory Rate | Continuously throughout 30 minute volunteer study
  Compared respiratory rate against capnometry.
Oxygen Saturation | Continuously throughout 30 minute volunteer study
  Did the novel system increase oxygen saturation?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Chanques G, Constantin JM, Sauter M, Jung B, Sebbane M, Verzilli D, Lefrant JY, Jaber S. Discomfort associated with underhumidified high-flow oxygen therapy in critically ill patients. Intensive Care Med. 2009 Jun;35(6):996-1003. doi: 10.1007/s00134-009-1456-x. Epub 2009 Mar 18. PMID 19294365
- [Background] Sasaki H, Yamakage M, Iwasaki S, Mizuuchi M, Namiki A. Design of oxygen delivery systems influences both effectiveness and comfort in adult volunteers. Can J Anaesth. 2003 Dec;50(10):1052-5. doi: 10.1007/BF03018373. PMID 14656787
- [Derived] Burk KM, Sakata DJ, Kuck K, Orr JA. Comparing Nasal End-Tidal Carbon Dioxide Measurement Variation and Agreement While Delivering Pulsed and Continuous Flow Oxygen in Volunteers and Patients. Anesth Analg. 2020 Mar;130(3):715-724. doi: 10.1213/ANE.0000000000004004. PMID 30633057